CLINICAL TRIAL: NCT05445466
Title: Causal Lesion Network Guided Treatment of Bipolar Mania With Transcranial Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Paulo Lizano, Assistant Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022P000295
Record Dates: First submitted 2022-06-17; First posted 2022-07-06 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Bipolar Disorder; Schizo Affective Disorder
Keywords: Brain Stimulation; Mania
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders; Mania

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- HD-tDCS (Active Comparator): HD-tDCS; Two, twenty-minute sessions of tDCS to the OFC for 5 days (10 total sessions)
  Interventions: Device: High-Definition Transcranial Electrical-Current Stimulation
- HD-tACS (alpha, 10 Hz) (Active Comparator): 10 Hz HD-tACS; Two, twenty-minute sessions of tACS to the OFC for 5 days (10 total sessions).
  Interventions: Device: High-Definition Transcranial Alternate-Current Stimulation
- Personalized Beta-Gamma HD-tACS (Active Comparator): Personalized HD-tACS; Two, twenty-minute sessions of tACS to the OFC for 5 days (10 total sessions).
  Interventions: Device: High-Definition Personalized Beta-Gamma Electrical Stimulation

INTERVENTIONS:
Device: High-Definition Transcranial Electrical-Current Stimulation — Non-frequency dependent transcranial electrical stimulation condition for 5 days of twice a day treatment
  Other Names: Soterix Medical; GTEN 200
  Arms: HD-tDCS
Device: High-Definition Transcranial Alternate-Current Stimulation — Active-control stimulation condition will target alpha (10 Hz) for 5 days of twice a day treatment
  Other Names: Soterix Medical; GTEN 200
  Arms: HD-tACS (alpha, 10 Hz)
Device: High-Definition Personalized Beta-Gamma Electrical Stimulation — Personalized beta-gamma electrical stimulation for 5 days of twice a day treatment
  Other Names: Soterix Medical; GTEN 200
  Arms: Personalized Beta-Gamma HD-tACS

SUMMARY:
Mania is a core symptom of bipolar disorder involving periods of euphoria. Decreased inhibitory control, increased risk-taking behaviors, and aberrant reward processing are some of the more recognized symptoms of bipolar disorder and are included in the diagnostic criteria for mania. Current drug therapies for mania are frequently intolerable, ineffective, and carry significant risk for side effects. Presently there are no neurobiologically informed therapies that treat or prevent mania. However, using a newly validated technique termed lesion network mapping, researchers demonstrated that focal brain lesions having a causal role in the development of mania in people without a psychiatric history can occur in different brain locations, such as the right orbitofrontal cortex (OFC), right dorsolateral prefrontal cortex (DLPFC), and right inferior temporal gyrus (ITG). This lesion network evidence converges with existing cross-sectional and longitudinal observations in bipolar mania that have identified specific disruptions in network communication between the amygdala and ventro-lateral prefrontal cortex. The OFC is associated with inhibitory control, risk-taking behavior, and reward learning which are major components of bipolar mania. Thus, the association between OFC with mania symptoms, inhibitory control, risk-taking behavior, and reward processing suggests that this region could be targeted using non-invasive brain stimulation.

DETAILED DESCRIPTION:
Mania is a core symptom of bipolar disorder involving periods of euphoria, delusions, and overactivity. Mania occurs in multiple medical and psychiatric illnesses and can be refractory to existing treatments. Two recent studies using brain lesion mapping of psychiatrically healthy individuals presenting with mania identified causal locations in the brain, including the orbitofrontal cortex (OFC), dorsolateral prefrontal cortex (DLPFC), and inferior temporal gyrus (ITG), that were associated with new onset mania symptoms. Moreover, these identified brain regions have also been implicated in bipolar mania with specific disruption in network communication between the amygdala and ventro-lateral prefrontal cortex. The OFC is of particular interest because it is a brain structure that is associated with inhibitory control, risk-taking behavior and reward, which are major behavioral components of mania. Thus, the association between OFC with mania symptoms, inhibitory control, risk-taking behavior and reward suggests that this region could be targeted using noninvasive brain stimulation. While several studies have non-invasively targeted the DLPFC for mania, no study to date has non-invasively stimulated the OFC with either transcranial direct current stimulation (tDCS) or alternating current (tACS) in bipolar disorder and examined its effects on mania, inhibitory control, or risk-taking behavior. However, a study in healthy volunteers showed that cathodal stimulation to the OFC enhanced inhibitory control and decreased risk-taking behavior. Recently, researches have showed that targeting the OFC with tACS, personalized to the individual's intrinsic beta-gamma frequency of the reward network, that individuals showed rapid, reversible, frequency-specific modulation of reward-guided choice behavior and learning. Here we aim to answer the question of whether noninvasive brain stimulation when optimally targeted and personalized to an individual's beta-gamma frequency to the OFC can improve emotional cognitive processing and mania symptoms compared to tDCS or sham targeting. The knowledge gained from this study will provide a marker for clinical response and allow personalized treatment for patients with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years of age
2. Proficient in English
3. Able to give informed consent
4. Meet diagnostic criteria for bipolar disorder or schizoaffective disorder, bipolar type as verified by the SCID
5. History of mania ( >1 lifetime episode)
6. Experiencing mild to moderate symptoms of mania
7. No changes to mood stabilizing medications for a period of 2 weeks prior to participation
8. Has not recently participated in tES/TMS treatments

Exclusion Criteria:

1. Substance abuse or dependence (w/in past 6 months)
2. Those who are pregnant/breastfeeding
3. History of head injury with > 15 minutes of loss of consciousness/mal sequelae
4. DSM-V intellectual disability
5. Having a non-removable ferromagnetic metal within the body (particularly in the head)
6. History of seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Lizano, MD,PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Individuals were randomized into 1 of 3 protocol arms (tDCS, 10hz tACS or personalized tACS)
Groups:
- HD-tACS (Alpha, 10 Hz): 10 Hz HD-tACS; Two, twenty-minute sessions of tACS to the OFC for 5 days (10 total sessions).
  High-Definition Transcranial Alternate-Current Stimulation: 10hz HD-tACS stimulation condition will target alpha (10 Hz) for 5 days of twice a day treatment.
Period: Overall Study
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma HD-tACS
Started | 5 | 4 | 5
Day 5 | 5 | 4 | 5
1 Month | 5 | 4 | 5
3 Month | 3 | 2 | 4
Completed | 3 | 2 | 4
Not Completed | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- HD-tACS (Alpha, 10 Hz): 10 Hz HD-tACS; Two, twenty-minute sessions of passive sham control to the OFC for a 30 second ramped up and down at the beginning and end of the 20 min period for 5 days (10 total sessions).
  High-Definition Transcranial Alternate-Current Stimulation: Active-control stimulation condition will target alpha (10 Hz) for 5 days of twice a day treatment
- Personalized Beta-Gamma HD-tACS: Personalized HD-tACS; Two, twenty-minute sessions of tACS to the OFC for 5 days (10 total sessions).
  High-Definition Personalized Transcranial (Beta-Gamma) Electrical Stimulation: Personalized beta-gamma electrical stimulation for 5 days of twice a day treatment
- Total: Total of all reporting groups
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma HD-tACS | Total
Number analyzed (Participants) | 5 | 4 | 5 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 5 | 14
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (10.402) | 38.25 (12.685) | 30.2 (11.476) | 34.29 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 7
  Male | 2 | 2 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 5 | 4 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 5 | 14
Altman Self-Rating Mania Scale (ASRM) [Median (Inter-Quartile Range); unit: score on a scale] — The ASRM is a 5-item self rating mania scale, assessing the presence and severity of manic symptoms. The scores for all five items are added together, resulting in a total score that can range from 0 to 20. A score of 6 or higher indicates a high probability of a manic or hypomanic condition.
  score on a scale | 5 [4 to 5] | 7 [3.75 to 9.5] | 3 [3 to 5] | 5 [3 to 7.25]

OUTCOME MEASURES:

1. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: Measuring total Mania scores; 11 items used to access severity of mania (total score 0-60); higher scores represent higher severity of symptoms
Time Frame: Change from baseline to 5 Day follow-up
Population: Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Personalized Beta-Gamma tACS: Personalized HD-tACS; Two, twenty-minute sessions of tACS to the OFC for 5 days (10 total sessions).
  High-Definition Personalized Transcranial (Beta-Gamma) Electrical Stimulation: Personalized beta-gamma electrical stimulation for 5 days of twice a day treatment
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 5.5 [0.5 to 6] | 11.8 [9.575 to 13.25] | 7.5 [5.5 to 8]
  Day 5 | 3 [2 to 3.5] | 8 [4.75 to 11.125] | 3 [1.5 to 13]

2. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: as for outcome 1
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice" R package used for 1 individual 1 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 5.5 [0.5 to 6] | 11.8 [9.575 to 13.25] | 7.5 [5.5 to 8]
  1 Month | 1.5 [1.5 to 4] | 11 [8 to 14.25] | 4 [1.5 to 5.5]

3. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: as for outcome 1
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R package used to impute 5 individuals 3 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 5.5 [0.5 to 6] | 11.8 [9.575 to 13.25] | 7.5 [5.5 to 8]
  3 Month | 2.6 [1.5 to 3.5] | 7.5 [5 to 9.625] | 2 [0.5 to 7]

4. Primary Outcome: Altman Self-Rating Mania Scale (ASRM)
Description: The ASRM is a 5-item self rating mania scale, assessing the presence and severity of manic symptoms. The scores for all five items are added together, resulting in a total score that can range from 0 to 20. A score of 6 or higher indicates a high probability of a manic or hypomanic condition.
Time Frame: Change from baseline to 5 Day follow-up
Population: Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 5 [4 to 5] | 7 [3.75 to 9.5] | 3 [3 to 5]
  Day 5 | 7 [4 to 8] | 2 [1 to 4.25] | 5 [5 to 7]

5. Primary Outcome: Altman Self-Rating Mania Scale (ASRM)
Description: as for outcome 4
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice' R package used to impute 1 individual's 1 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 5 [4 to 5] | 7 [3.75 to 9.5] | 3 [3 to 5]
  1 Month | 2 [1 to 3] | 4 [2.25 to 6.25] | 5 [5 to 6]

6. Primary Outcome: Altman Self-Rating Mania Scale (ASRM)
Description: as for outcome 4
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R package used to impute 5 individuals 3 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 5 [4 to 5] | 7 [3.75 to 9.5] | 3 [3 to 5]
  3 Month | 2 [2 to 4] | 3.6 [2.25 to 4.5] | 6 [5 to 7.2]

7. Primary Outcome: Psychiatric Hospitalizations for Mania Post Study Entry
Description: Psychiatric hospitalization for mania. Count of hospitalizations from baseline to end of study period assessed at Day 5, 1 Month & 3 Month.
Time Frame: Cumulative count of hospitalizations for mania from baseline to end of study
Population: Cumulative count of hospitalizations for mania from baseline to end of study
Measure: Number; unit: number of hospitalizations
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
number of hospitalizations
  Baseline | 0 | 0 | 0
  Day 5 | 0 | 0 | 0
  1 Month | 0 | 1 | 0
  3 Month | 0 | 0 | 0

8. Secondary Outcome: Balloon Analogue Risk Task (BART)
Description: The BART is a computerized task the measures risk-taking behavior. Participants are tasked with inflating the virtual balloon. The number of pumps a participant chooses to make on each balloon is used as a measure of their risk-taking behavior. More pumps generally indicate a higher tolerance for risk. The balloon bursts at a given point if the participant overfills it. Number of popped balloons reported for a given trial.
Time Frame: Change from baseline to 5 Day follow-up
Measure: Median (Inter-Quartile Range); unit: popped balloons
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
popped balloons
  Baseline | 16 [10 to 17] | 13.5 [11.5 to 15.25] | 13 [11 to 19]
  Day 5 | 17 [16 to 17] | 13.5 [7.75 to 20] | 18 [14 to 25]

9. Secondary Outcome: Balloon Analogue Risk Task (BART)
Description: as for outcome 8
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice' R package used to impute 1 individual's 1 Month data
Measure: Median (Inter-Quartile Range); unit: popped balloons
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
popped balloons
  Baseline | 16 [10 to 17] | 13.5 [11.5 to 15.25] | 13 [11 to 19]
  1 Month | 15 [15 to 16] | 14.1 [10.5 to 18.65] | 27 [17 to 28]

10. Secondary Outcome: Balloon Analogue Risk Task (BART)
Description: as for outcome 8
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R packaged used to impute 5 individuals' 3 Month data
Measure: Median (Inter-Quartile Range); unit: popped balloons
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
popped balloons
  Baseline | 16 [10 to 17] | 13.5 [11.5 to 15.25] | 13 [11 to 19]
  3 Month | 12.2 [11 to 14] | 14.7 [11.75 to 18.3] | 18 [14 to 22]

11. Secondary Outcome: The Go/No Go Task
Description: The Go/No Go Task is a computerized task that measures impulsiveness. Participants presented with Go (to respond) and no Go (when not to respond) instructions. Two trials are performed. The first trial consist of two distinct auditory stimuli (both Go stimuli) where the participant is asked to respond with a different number of mouse clicks to the stimuli respectively. The second trial, has a no Go stimuli (where the participant is suppose to withhold a response) and a go stimuli. Reaction time for correct trials only for the entire task are reported in milliseconds.
Time Frame: Change from baseline to 5 Day follow-up
Measure: Median (Inter-Quartile Range); unit: reaction time (ms) on task
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
reaction time (ms) on task
  Baseline | 876.9768638 [675.4974359 to 923.1895604] | 954.3716154 [894.5683204 to 964.7482317] | 859.6685714 [857.6372796 to 1139.709184]
  Day 5 | 927.1679389 [925.6649616 to 1011.031746] | 878.0193364 [871.9321033 to 915.1828861] | 917.7871795 [805.0713097 to 994.2446809]

12. Secondary Outcome: The Go/No Go Task
Description: as for outcome 11
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice' R package used for 1 individual's 1 Month data
Measure: Median (Inter-Quartile Range); unit: reaction time (ms) on task
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
reaction time (ms) on task
  Baseline | 876.9768638 [675.4974359 to 923.1895604] | 954.3716154 [894.5683204 to 964.7482317] | 859.6685714 [857.6372796 to 1139.709184]
  1 Month | 923.5850515 [914.8220551 to 939.1815857] | 919.8986144 [910.2266457 to 942.2465073] | 880.3450882 [838.5765306 to 993.5419847]

13. Secondary Outcome: The Go/No Go Task
Description: as for outcome 11
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R package used to impute 5 individuals 3 Month data
Measure: Median (Inter-Quartile Range); unit: reaction time (ms) on task
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
reaction time (ms) on task
  Baseline | 876.9768638 [675.4974359 to 923.1895604] | 954.3716154 [894.5683204 to 964.7482317] | 859.6685714 [857.6372796 to 1139.709184]
  3 Month | 931.8461538 [902.5325077 to 953.3693886] | 925.0182573 [897.7525324 to 951.0867497] | 845.64 [803.9641944 to 930.8737113]

14. Secondary Outcome: Electroencephalography (EEG) Resting State
Description: Measuring neural activity at rest consisting of 5 minutes of eyes-open resting-state EEG (rsEEG) was recorded. Fast Fourier transformations were conducted on data, resulting in 4 frequency bands: delta/theta, alpha, beta, and gamma.
Time Frame: Change from baseline to 5 Day follow-up
Population: Delta/Theta represents the range of 2-7Hz
Measure: Median (Inter-Quartile Range); unit: peak amplitude measured in microvolts
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
peak amplitude measured in microvolts
  Baseline Delta/Theta | -9.261 [-9.654 to -8.720] | -7.555 [-8.544 to -4.817] | -6.410 [-9.009 to -5.245]
  Baseline Alpha | -13.336 [-13.435 to -12.118] | -8.834 [-9.639 to -6.513] | -11.185 [-12.112 to -6.792]
  Baseline Beta | -17.191 [-18.932 to -17.076] | -11.636 [-13.139 to -10.309] | -17.344 [-18.287 to -16.151]
  Baseline Gamma | -21.651 [-23.656 to -20.064] | -17.087 [-18.618 to -15.387] | -24.011 [-24.143 to -20.892]
  Day 5 Delta/Theta | -8.844 [-10.331 to -8.711] | -3.373 [-4.858 to -1.851] | -3.567 [-8.164 to -3.369]
  Day 5 Alpha | -12.946 [-14.470 to -11.370] | -8.241 [-9.049 to -6.130] | -8.445 [-12.857 to -6.938]
  Day 5 Beta | -17.898 [-17.968 to -16.311] | -12.266 [-13.787 to -10.604] | -16.360 [-16.494 to -16.166]
  Day 5 Gamma | -20.695 [-22.511 to -20.690] | -16.232 [-18.035 to -15.364] | -22.996 [-24.261 to -22.019]

15. Secondary Outcome: Electroencephalography (EEG) Resting State
Description: as for outcome 14
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice' R package used to impute 1 individual's 1 Month Data. Delta/Theta represents the range of 2-7Hz.
Measure: Median (Inter-Quartile Range); unit: peak amplitude measured in microvolts
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
peak amplitude measured in microvolts
  Baseline Delta/Theta | -9.261 [-9.654 to -8.720] | -7.555 [-8.544 to -4.817] | -6.410 [-9.009 to -5.245]
  Baseline Alpha | -13.336 [-13.435 to -12.118] | -8.834 [-9.639 to -6.513] | -11.185 [-12.112 to -6.792]
  Baseline Beta | -17.191 [-18.932 to -17.076] | -11.636 [-13.139 to -10.309] | -17.344 [-18.287 to -16.151]
  Baseline Gamma | -21.651 [-23.656 to -20.064] | -17.087 [-18.618 to -15.387] | -24.011 [-24.143 to -20.892]
  1 Month Delta/Theta | -9.775 [-10.242 to -8.359] | -8.373 [-9.455 to -7.109] | -4.015 [-8.554 to -3.696]
  1 Month Alpha | -14.921 [-15.199 to -11.276] | -11.520 [-12.060 to -10.555] | -10.646 [-12.675 to -7.025]
  1 Month Beta | -16.627 [-17.518 to -16.425] | -13.489 [-14.057 to -13.213] | -17.502 [-18.891 to -16.455]
  1 Month Gamma | -19.358 [-19.363 to -19.102] | -19.739 [-21.221 to -18.424] | -22.594 [-24.795 to -21.966]

16. Secondary Outcome: Electroencephalography (EEG) Resting State
Description: as for outcome 14
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R package used to impute 5 individuals 3 Month data. Delta/Theta represents the range of 2-7Hz.
Measure: Median (Inter-Quartile Range); unit: peak amplitude measured in microvolts
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
peak amplitude measured in microvolts
  Baseline Delta/Theta | -9.261 [-9.654 to -8.720] | -7.555 [-8.544 to -4.817] | -6.410 [-9.009 to -5.245]
  Baseline Alpha | -13.336 [-13.435 to -12.118] | -8.834 [-9.639 to -6.513] | -11.185 [-12.112 to -6.792]
  Baseline Beta | -17.191 [-18.932 to -17.076] | -11.636 [-13.139 to -10.309] | -17.344 [-18.287 to -16.151]
  Baseline Gamma | -21.651 [-23.656 to -20.064] | -17.087 [-18.618 to -15.387] | -24.011 [-24.143 to -20.892]
  3 Month Delta/Theta | -8.764 [-9.704 to -8.220] | -7.362 [-8.040 to -6.876] | -3.686 [-8.560 to -3.538]
  3 Month Alpha | -14.041 [-14.599 to -12.839] | -10.615 [-10.914 to -9.682] | -7.918 [-11.435 to -7.331]
  3 Month Beta | -17.323 [-18.195 to -17.186] | -13.074 [-13.410 to -12.645] | -17.643 [-18.436 to -16.060]
  3 Month Gamma | -21.479 [-21.743 to -20.864] | -19.348 [-20.173 to -17.743] | -23.863 [-24.238 to -23.257]

17. Secondary Outcome: Reinforcement Learning Task
Description: The reinforcement learning task is a monetary based learning tasks that included reward and punishment trails. The task presents multiple trials of stimuli where the participant chooses 1 of 2 stimuli presented at a time (one of which is associated with punishment represented by loss of monetary reward while the other is associated with gain of monetary reward). EEG is record during the task and signal is captured during the participants choose and the feedback received. Reported is the peak beta/gamma range response derived from the EEG during reward feedback. This measurement is used from the baseline assessment to inform the personalized beta-gamma range stimulation for the Personalized Beta-Gamma tACS group.
Time Frame: Change from baseline to 5 Day follow-up
Measure: Median (Inter-Quartile Range); unit: peak frequency measured in hertz
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
peak frequency measured in hertz
  Baseline | 26 [23.5 to 29] | 25.25 [20 to 30.875] | 32 [31 to 32]
  Day 5 | 28.5 [25 to 30.5] | 33.75 [30.5 to 35] | 22 [22 to 35]

18. Secondary Outcome: Reinforcement Learning Task
Description: as for outcome 17
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice' R package used to impute 1 individual's 1 Month data
Measure: Median (Inter-Quartile Range); unit: peak frequency measured in hertz
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
peak frequency measured in hertz
  Baseline | 26 [23.5 to 29] | 25.25 [20 to 30.875] | 32 [31 to 32]
  1 Month | 25 [21.5 to 30.5] | 28.75 [28.5 to 29.875] | 27.5 [22.5 to 28.5]

19. Secondary Outcome: Reinforcement Learning Task
Description: as for outcome 17
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R package used for imputing 5 individuals 3 Month data
Measure: Median (Inter-Quartile Range); unit: peak frequency measured in hertz
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
peak frequency measured in hertz
  Baseline | 26 [23.5 to 29] | 25.25 [20 to 30.875] | 32 [31 to 32]
  3 Month | 25.5 [23.7 to 25.6] | 29.25 [28.625 to 29.5] | 27.5 [27 to 30]

20. Secondary Outcome: Social Functioning Scale (SFS)
Description: The SFS a self-report questionnaire initially designed for people diagnosed with Schizophrenia; consists of 79 items designed to reflect the social skills and performances in different areas of life. Subscores are summed together for a total score. Total score of SFS ranges between 0-223 points. Higher scores mean better social functioning.
Time Frame: Change from baseline to 5 Day follow-up
Population: Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 161 [133 to 166] | 125.5 [120 to 129.25] | 142 [129 to 152]
  Day 5 | 159 [138.4 to 159.4] | 125.7 [123.95 to 128.05] | 144 [124.2 to 145.4]

21. Secondary Outcome: Social Functioning Scale (SFS)
Description: as for outcome 20
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice' R package used to impute 1 individual's 1 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 161 [133 to 166] | 125.5 [120 to 129.25] | 142 [129 to 152]
  1 Month | 160 [133 to 171] | 130.5 [122 to 139] | 134 [131 to 145]

22. Secondary Outcome: Social Functioning Scale (SFS)
Description: as for outcome 20
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R package used to impute 5 individuals 3 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 161 [133 to 166] | 125.5 [120 to 129.25] | 142 [129 to 152]
  3 Month | 156.6 [134 to 164] | 127.2 [116.75 to 135.75] | 150 [135 to 170]

23. Secondary Outcome: Global Assessment of Functioning (GAF)
Description: The GAF measures how symptoms affect individuals day-to-day life; scored from 0 to 100
Time Frame: Change from baseline to 5 Day follow-up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 65 [60 to 65] | 46 [40.75 to 53.25] | 59 [51 to 60]
  Day 5 | 61 [61 to 61] | 50.5 [48.75 to 52] | 60 [57 to 60]

24. Secondary Outcome: Global Assessment of Functioning (GAF)
Description: The GAF measures how symptoms affect individuals day-to-day life; scored from 0 to 100
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice' R package used to impute 1 individual's 1 Month data
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 65 [60 to 65] | 46 [40.75 to 53.25] | 59 [51 to 60]
  1 Month | 67 [65 to 70] | 51 [50.75 to 51.25] | 55 [55 to 60]

25. Secondary Outcome: Global Assessment of Functioning (GAF)
Description: The GAF measures how symptoms affect individuals day-to-day life; scored from 0 to 100
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R package used to impute 5 individuals 3 Month data
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 65 [60 to 65] | 46 [40.75 to 53.25] | 59 [51 to 60]
  3 Month | 65 [65 to 67] | 52.1 [50.55 to 53.65] | 61 [60 to 61]

26. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: 30 items included in the PANSS measuring positive, negative and general symptoms; 7 related to positive symptoms, 7 for negative symptoms, and 16 for general psychopathology Scale. Ranges are 7 to 49 for the Positive and Negative Scales, and 16 to 112 for the General Psychopathology Scale. Scores summed for Total Score on scale (30 to 210). Higher scores mean worse clinical symptoms. Total score reported.
Time Frame: Change from baseline to 5 Day follow-up
Population: Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 49 [49 to 55] | 71 [60.75 to 78.5] | 68 [61 to 69]
  Day 5 | 52 [48 to 56] | 74.5 [69 to 77] | 56 [49 to 68]

27. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: as for outcome 26
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice' R package used to impute 1 individuals 1 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 49 [49 to 55] | 71 [60.75 to 78.5] | 68 [61 to 69]
  1 Month | 50 [42 to 54] | 75 [73.5 to 78] | 55 [52 to 55]

28. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: as for outcome 26
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R package used to impute 5 individuals 3 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 49 [49 to 55] | 71 [60.75 to 78.5] | 68 [61 to 69]
  3 Month | 54.8 [48.6 to 55] | 73.3 [72.25 to 77.45] | 52 [51 to 54.6]

29. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: The MADRS is designed to measure depression and severity of symptoms; 0 to 6 indicates no depression, 7 to 19 indicates mild depression, 20 to 34 indicates moderate depression, 35 and greater indicates severe depression. Total score reported (0 to 60).
Time Frame: Change from baseline to 5 Day follow-up
Population: Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 8 [8 to 11] | 17.5 [11.5 to 23.75] | 10 [8 to 29]
  Day 5 | 7 [6 to 13] | 14.5 [12 to 16] | 7 [7 to 10]

30. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: as for outcome 29
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice' R package used to impute 1 individual's 1 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 8 [8 to 11] | 17.5 [11.5 to 23.75] | 10 [8 to 29]
  1 Month | 7 [6 to 13] | 16 [15.75 to 17.5] | 8 [5 to 8]

31. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: as for outcome 29
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R package used to impute 5 individuals 3 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 8 [8 to 11] | 17.5 [11.5 to 23.75] | 10 [8 to 29]
  3 Month | 8 [5 to 8] | 19.2 [16.25 to 26] | 6 [6 to 9]

32. Secondary Outcome: Barratt Impulsiveness Scale-11 (BIS-11)
Description: The BIS-11 is designed to assess the personality/behavioral impulsiveness. The BIS-11 has 30 items and is scored appropriately. Scored to yield a total score, three second-order factors, and six first-order factors. Each question has a 4-point scale ranging from 1 (rarely/never) to 4 (almost always/always). Higher scores mean more impulsive behavior. Total score reported (30-120).
Time Frame: Change from baseline to 5 Day follow-up
Population: Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 37 [36 to 41] | 35 [29 to 41.75] | 42 [40 to 42]
  Day 5 | 38 [36 to 41] | 38.5 [35.5 to 43] | 41 [32 to 44]

33. Secondary Outcome: Barratt Impulsiveness Scale-11 (BIS-11)
Description: as for outcome 32
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice' R package used to impute 1 individual's 1 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 37 [36 to 41] | 35 [29 to 41.75] | 42 [40 to 42]
  1 Month | 35 [34 to 40] | 38 [27.5 to 47.25] | 40 [36 to 42]

34. Secondary Outcome: Barratt Impulsiveness Scale-11 (BIS-11)
Description: as for outcome 32
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R package used to impute 5 individuals 3 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a scale
  Baseline | 37 [36 to 41] | 35 [29 to 41.75] | 42 [40 to 42]
  3 Month | 35.2 [31 to 35.6] | 38 [37 to 38.15] | 36 [35.2 to 36]

35. Secondary Outcome: Brief Assessment of Cognition (BACS)
Description: The BACS is designed to assess several domains of cognition; Verbal Memory; Processing Speed; Working Memory; Verbal Fluency; Motor Function; Executive Functioning. Higher scores indicate better cognitive functioning. Total score reported after being transformed into z score based on normative scoring provide by test makers.
Time Frame: Change from baseline to 5 Day follow-up
Population: Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a test
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a test
  Baseline | 0.44 [-0.79 to 0.71] | -0.66 [-1.065 to 0.0025] | 0.25 [-0.35 to 0.76]
  Day 5 | 0.43 [-0.26 to 0.71] | -0.74 [-0.97 to -0.3525] | 0.3 [0.21 to 0.77]

36. Secondary Outcome: Brief Assessment of Cognition (BACS)
Description: as for outcome 35
Time Frame: Change from baseline to 1-month follow-up
Population: 'Mice' R package used to impute 1 individual's 1 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a test
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a test
  Baseline | 0.44 [-0.79 to 0.71] | -0.66 [-1.065 to 0.0025] | 0.25 [-0.35 to 0.76]
  1 Month | 0.01 [-0.07 to 0.51] | -1.26 [-1.3975 to -0.9485] | 0.74 [-0.09 to 0.9]

37. Secondary Outcome: Brief Assessment of Cognition (BACS)
Description: as for outcome 35
Time Frame: Change from baseline to 3-month follow-up
Population: 'Mice' R package used to impute 5 individuals 3 Month data. Total score reported.
Measure: Median (Inter-Quartile Range); unit: score on a test
Arm/Group | HD-tDCS | HD-tACS (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
Number analyzed (Participants) | 5 | 4 | 5
score on a test
  Baseline | 0.44 [-0.79 to 0.71] | -0.66 [-1.065 to 0.0025] | 0.25 [-0.35 to 0.76]
  3 Month | 0.18 [-0.146 to 0.44] | -0.602 [-0.7055 to -0.456] | 0.97 [0.384 to 1.58]

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 3 months after tES treatment (10 sessions over 1 week) was completed.
Groups:
- Active HD-tDCS: tDCS; Two, twenty-minute sessions of tDCS to the OFC for 5 days (10 total sessions).
  High-Definition Transcranial Electrical-Current Stimulation: Non-frequency dependent transcranial electrical stimulation condition for 5 days of twice a day treatment
- Active Control (Alpha, 10 Hz): Passive sham control; Two, twenty-minute sessions of passive sham control to the OFC for a 30 second ramped up and down at the beginning and end of the 20 min period for 5 days (10 total sessions).
  High-Definition Transcranial Alternate-Current Stimulation: Active-control stimulation condition will target alpha (10 Hz) for 5 days of twice a day treatment
- Personalized Beta-Gamma tACS: tACS; Two, twenty-minute sessions of tACS to the OFC for 5 days (10 total sessions).
  High-Definition Personalized Beta-Gamma Electrical Stimulation: Personalized beta-gamma electrical stimulation for 5 days of twice a day treatment
Arm/Group | Active HD-tDCS | Active Control (Alpha, 10 Hz) | Personalized Beta-Gamma tACS
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 0/4 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active HD-tDCS (N=5) | Active Control (Alpha, 10 Hz) (N=4) | Personalized Beta-Gamma tACS (N=5)
Eye Fatigue/Pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — Individual reported eye pain/fatigue after completing 10 sessions of stimulation. The individual was suffering from a common cold at the time. Symptoms resolved on their own after a few days.

LIMITATIONS AND CAVEATS:
Overall recruitment numbers were low which led to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT05445466/Prot_SAP_000.pdf